CLINICAL TRIAL: NCT06383728
Title: Osimertinib as Neoadjuvant Therapy in Patients With Resectable Stage II-IIIB EGFR-mutated Lung Squamous Cell Carcinoma: A Single-centre, Single-arm, Phase 2 Trial
Brief Title: Neoadjuvant Targeted Therapy in Patients With Resectable EGFR-mutated Lung Squamous Cell Carcinoma
Acronym: GALAXY-02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Shuben Li, Deputy Administrative Director of thoracic surgery, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES-2024-014-02
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer; Carcinoma, Squamous Cell
Keywords: neoadjuvant targeted therapy; EGFR-mutated lung squamous cell carcinoma; surgery
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Squamous Cell | interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: Patients with resectable stage II-IIIB EGFR-mutated lung squamous cell carcinoma receive osimertinib (80mg/d, ≥9 weeks)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib (Experimental): Patients with resectable stage II-IIIB EGFR-mutated lung squamous cell carcinoma will receive Osimertinib ( 80mg/d, ≥9 weeks).
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Patients with resectable stage II-IIIB EGFR-mutated lung squamous cell carcinoma will receive Osimertinib ( 80mg/d, ≥9 weeks).
  Other Names: Tagrisso

SUMMARY:
Previous trials, such as ADURA and CTONG, have demonstrated the benefits of neoadjuvant targeted therapy in patient with EGFR mutations , which can effectively reduce the extent of tumors and improve the survival outcomes. However, clinical trials of neoadjuvant targeted therapy in NSCLC have rarely enrolled patients with EGFR-mutated lung squamous cell carcinoma due to its rarity, which means that the safety and feasibility of neoadjuvant osimertinib in patients with resectable stage II-IIIB EGFR-mutated lung squamous cell carcinoma remains controversial.

DETAILED DESCRIPTION:
This trial aims to investigated the safety and feasibility of neoadjuvant osimertinib in patients with resectable stage II-IIIB EGFR-mutated lung squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Chest CT and pathological examination confirmed as resectable II-IIIB lung squamous cell carcinoma;
2. Gene text confirmed EGFR mutation;
3. PET-CT confirmed no metastasis;
4. ECOG physical status score 0-1;
5. Age ≥ 18 years;
6. Have one measurable lesion at least;
7. Good function of other major organs (liver, kidney, blood system, etc.):-absolute neutrophil count ((ANC) ≥ 1.5 × 109), platelet (≥ 100 × 109), hemoglobin (≥ 90g/L). Note: patients shall not receive blood transfusion or growth factor support within 14 days before blood collection during the screening period;-International standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 × normal upper limit (ULN);-activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;- serum total bilirubin ≤ 1.5 × ULN (Gilbert syndrome patients with total bilirubin must be < 3×ULN). Fertile female patients with aspartate and alanine aminotransferase (AST and ALT) ≤ 2.5 × ULN, or liver metastasis with AST and ALT ≤ 5 × ULN
8. Fertile female patients must voluntarily take effective contraceptive measures more than 120 days after treatment, and the urine or serum pregnancy test results less than 7 days before entering the group were negative. Unsterilized male patients must voluntarily take effective contraceptive measures ≥ 120 days after treatment;
9. Sign informed consent.

Exclusion Criteria:

1. Patients with other malignant tumors in the five years before the start of this trial.
2. Complicated with unstable systemic diseases, including active infections, uncontrolled hypertension, unstable angina pectoris, congestive heart failure [higher than II (New York College of Cardiology)], severe arrhythmias, liver, kidney or metabolic diseases;
3. Active, known or suspected autoimmune diseases, or autoimmune paraneoplastic syndrome requiring systemic treatment;
4. A history of active bleeding or embolism within 6 months, or received thrombolysis or anticoagulation therapy, or the researchers believe that there is an obvious tendency of gastrointestinal bleeding (such as esophageal varices have the risk of bleeding, local active ulcer lesions, etc.);
5. Allergic to experimental drugs;
6. Complicated with HIV infection or active hepatitis.
7. Vaccination within 4 weeks before the start of this trial;
8. Those who had undergone other major operations or severe injuries within the previous 2 months;
9. Clinically uncontrolled pleural effusion or ascites requiring pleural or abdominal puncture drainage within 2 weeks before admission;
10. Pregnant or lactating women;
11. Those with neurological diseases or mental disorders;
12. Participated in another therapeutic clinical study at the same time;
13. Other researchers did not consider it appropriate to enroll in the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | analysis is completed 4 weeks after neoadjuvant treatment
  Defined as the proportion of participants who had a complete response (CR) or partial response (PR) according to RECIST version 1.1 after treatment.
Safety: frequency of severe adverse events | from the participants enrolling to 30 days after the last drug administration or 30 days after surgery.
  The frequency of severe adverse events from the participants enrolling to 30 days after the last drug administration or 30 days after surgery.

SECONDARY OUTCOMES:
Major pathologic response, MPR | analysis is completed 4 weeks after surgery
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery.
R0 rate | analysis is completed 4 weeks after surgery
  There were no visible tumors in the surgical margin, and the tumor cells in the surgical margin within 1mm were negative under the microscope.
Progression-free survival (PFS) | 2 years
  PFS is defined as the time from the enrollment of the subject to the first determination of disease progression or death of any cause according to RECISTv1.1, whichever occurs first.
Overall survival (OS) | 5 years
  It is defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date. In the event of a patient with the survival status unknown, the date when the patient is last known to be alive will be used for interpolation (censoring).
Disease control rate (DCR) | 2 years
  The proportion of patients whose best overall remission (BOR) is CR, PR or disease stable (SD) according to RECISTv1.1 evaluation
Duration of remission (DOR) | 2 years
  According to the time from the first recording of objective remission to relapse or death from any cause determined by RECISTv1.1, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: shuben Li, Doctor, Study Director — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No